CLINICAL TRIAL: NCT01837394
Title: Ultrasound-guided Block of the Saphenous Nerve and Obturator Nerve, Posterior Branch, for Postoperative Pain Management After Ambulatory Knee Arthroscopy
Brief Title: Ultrasound-guided Blocks for Ambulatory Knee Arthroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jens Borglum Neimann (Other)
Responsible Party: Sponsor-Investigator, Jens Borglum Neimann, MD, PhD, MBA, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-2-2011-029
Record Dates: First submitted 2013-04-15; First posted 2013-04-23 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Postoperative Pain; Postoperative Nausea and Vomiting; Postoperative Function Level
Keywords: Nerve block; Ultrasound; postoperative pain; Saphenous nerve; Obturator nerve
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Ropivacaine; Acetaminophen; Morphine; Ondansetron; Metoclopramide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Block arm (Active Comparator): Ultrasound guided block of the SN and ONP with 7.5 ml of Ropivacaine 7.5 mg/ml injected at each site, respectively, immediately prior to induction of general anesthesia. Standard postoperative analgesia with paracetamol 1 g every 6 hours and Morphine 5 mg as needed. Ondansetron or Metoclopramide as needed for nausea.
  Interventions: Procedure: Block of the SN and ONP; Drug: Paracetamol; Drug: Morphine; Drug: Ondansetron; Drug: Metoclopramide
- Placebo arm (Placebo Comparator): Ultrasound guided placebo block of the SN and ONP with 7.5 ml of isotonic saline solution injected at each site, respectively, immediately prior to induction of general anesthesia. Standard postoperative analgesia with paracetamol 1 g every 6 hours and Morphine 5 mg as needed. Ondansetron or Metoclopramide as needed for nausea.
  Interventions: Procedure: Placebo block; Drug: Paracetamol; Drug: Morphine; Drug: Ondansetron; Drug: Metoclopramide

INTERVENTIONS:
Procedure: Block of the SN and ONP — 7.5 ml of Ropivacaine 7.5 mg/ml injected at each site
  Other Names: Naropin
  Arms: Block arm
Procedure: Placebo block — 7.5 ml of isotonic saline solution 154 mmol/l injected at each site
  Other Names: NaCl
  Arms: Placebo arm
Drug: Paracetamol
  Other Names: Acetaminophen
Drug: Morphine — 5 mg as needed
Drug: Ondansetron — 4 mg i.v. as needed in the PACU
  Other Names: Zofran
Drug: Metoclopramide — 10 mg tablet as needed in the postoperative period after discharge from the PACU
  Other Names: Emperal; Primperan

SUMMARY:
In this study, we wish to investigate the effect of ultrasound (US) -guided block of the saphenous nerve (SN) and the posterior branch of the obturator nerve (ONP) on postoperative pain and the use of opioids (morphine-like pain medicine) in the first 24 hours following ambulatory knee arthroscopy.

We wish to investigate the analgesic effect of these two blocks compared to placebo (injection of local anesthetic with known pain blocking properties compared with injection of a saline solution), when used as a supplement to conventional oral analgesics.

We hypothesize that patients receiving the active treatment may experience less pain during the first 24 hours after their operation than patients receiving the placebo treatment, and possibly require less opioid analgesics, experience less opioid related side effects and have a higher function level in this period than patients receiving the placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

* Planned ambulatory knee arthroscopy, except cruciate ligament surgery
* American Society of Anesthesiologists (ASA) class 1-3

Exclusion Criteria:

* Cannot cooperate
* Do not speak or understand Danish
* Daily use of opioid analgesics
* Allergy towards any of the drugs used in the investigation
* Medicine abuse (at the investigators discretion)
* Alcohol abuse, as defined by the National Board of Health
* General anesthesia contraindicated, or the patient wants spinal anesthesia
* Visualization of necessary structures by ultrasound not possible, or block not possible for other technical reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Pain on knee flexion | 24 hours postoperatively
  VRS (Verbal Rating Scale) score 0-10 on active flexion of the knee to 45 degrees, measured at 0, ½, 1, 2, 3, 4, 6, 8, 12 and 24 hours postoperatively and analyzed by area under curve (AUC) analysis.

SECONDARY OUTCOMES:
Pain at rest | 24 hours postoperatively
  VRS (verbal rating score) 0-10 at rest, measured at 0, ½, 1, 2, 3, 4, 6, 8, 12 and 24 hours postoperatively and analyzed by area under curve (AUC) analysis.
Time to opioid intake | 24 hours postoperatively
  First time the patient needs to take supplementary opioids in the postoperative period
Total opioid intake | 24 hours
  Total dose of opioids taken in the first 24 hours postoperatively
Nausea | 24 hours postoperatively
  VRS score 0-10, measured at 0, ½, 1, 2, 3, 4, 6, 8, 12 and 24 hours postoperatively and analyzed by area under curve (AUC) analysis.
Vomiting | 24 hours
  Number of times the patient has vomited in the first 24 hours postoperatively.
Use of antiemetics | 24 hours
  Total dose of antiemetics taken during the first 24 hours postoperatively
PACU length of stay | 24 hours
  Total length of stay in the post anesthetic care unit (PACU) after the operation.
Function level: Barthel Index/100 | 24 hours
  Modified Barthel Index/100 score 24 hours after the operation.
Function level: Short form (SF) -8 | 24 hours
  Short form (SF) -8 questionnaire 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Bo Westergaard, MD, Principal Investigator — Department of Anesthesiology, Bispebjerg Hospital
Locations (1):
- Department of Anesthesiology, Bispebjerg Hospital, Copenhagen, Denmark